CLINICAL TRIAL: NCT05772312
Title: Quality of Life of Patients With Bone Tumors of the Lower Limbs Treated With Salvage Surgery: a Long-term Follow-up Study.
Brief Title: Quality of Life of Patients With Bone Tumor of the Lower Limbs Treated With Salvage Surgery
Acronym: Onco-QoL
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 5000
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Sarcoma, Ewing; Osteosarcoma; Bone Tumor
Keywords: quality of life; rehabilitation
MeSH Terms: conditions — Sarcoma, Ewing; Osteosarcoma; Bone Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to describe, through a minimum follow-up of 18 months, the quality of life of patients undergoing salvage surgery of lower limb for musculoskeletal tumors and to identify possible prognostic factor correlated.

Quality of life will be evaluated with Bt-DUX (Bt=bone tumor)

DETAILED DESCRIPTION:
Musculoskeletal cancers are extremely rare, accounting for approximately 0.2% of all cancers, 14% are bone sarcomas, which occur more frequently in children and adolescents. The most frequent location is at the metaphyseal level of the femur (42%) and tibia (19%).

Surgery and chemotherapy treatments have significantly increased survival rates for patients with bone tumor. Early rehabilitation of these patients after surgery is to promote recovery as early as possible with maximum autonomy. In literature, data about the association between the early functional recovery and quality of life are few. Long-term studies about the quality of life of these patients are so necessary. The quality of life is measured with several scale that included a set of non-specific domains for bone tumor patients. For this reason, a specific assessment scale was introduced and validated in 2013 to measure the quality of life of patients with bone cancer of the lower limbs, the Bt-DUX scale.

In 2019 the Bt-DUX scale was validated in Italian.

Considering the rarity of the disease, and verified that the number of patients treated in 2019 and 2020, is 30 and 32, respectively, the investigators estimate to enroll from January 2019 to June 2023 a number of patients equal to 100, considering a rejection rate of 10%.

Patient characteristics and scale values will be summarized using descriptive statistics (absolute frequencies and percentages for categorical variables, mean and standard deviation or median and interquartile range for continuous variables).

The variables collected will be: age, sex, diagnosis, type of surgery, site of tumour, complication (infection, relapses, metastasis), TESS (Toronto Extremity Salvage Score) (at 3 and 6 months), knee or hip flexion (at 3 and 6 months), quadriceps or hip abductor strength (at 3 and 6 months) and time up and go (at 3 and 6 months).

The relationship of patient characteristics with functional outcomes and quality of life will be investigated using multiple regression models, while the correlation between measures of functional recovery will be analyzed using Pearson's or Spearman's correlation coefficient, depending on the distribution of the variables considered.

The aim of the study is to describe the quality of life of patients undergoing salvage surgery of the lower limb for musculoskeletal tumors with a long follow-up and to investigate the association with early functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients 12 years of age or older with musculoskeletal cancer undergoing lower extremity salvage surgery

Exclusion Criteria:

* patients undergoing amputation
* patients with difficulties in understanding the Italian language

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with musculoskeletal tumor of the lower limbs who underwent salvage surgery at the "SC Clinica Ortopedica e Traumatologia III" of the Rizzoli Orthopedic Institute from January 2019 to June 2023 and will be followed up in the "SC Osteoncology, bone and soft tissues sarcomas and innovative therapies" of the same Institute for chemotherapy and physiotherapy treatment.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Bt-DUX scale | quality of life will be measured once in a time interval ranging from 18 months to 5 years post surgery
  The Bt-DUX scores reflect patients' personal impact: their individual values for cosmetic, social, emotional, and functional aspects of their life after surgery.
  The scoring of the items is done by abstract faces with varying expressions/smiley's, ranging from very happy (score 1) to sad (score 5). The raw item scores are converted into total and domain scores, ranging from 0 to 100, with the highest scores indicating better HRQoL (health related quality of life).

SECONDARY OUTCOMES:
TESS | TESS will be administered once in a time interval ranging from 18 months to 5 years post surgery
  The TESS is a self-administered questionnaire evaluating possible limitations in physical activity. A total of 30 questions are included in the TESS, and the degree of disability is rated from 0 (complete disability) to 5 (no functional impairment) in each item. Similar to MSTS (musculoskeletal tumour society score) for lower extremity, the final TESS score is converted to a score ranging from 0 to 100 points. If a question in TESS score does not apply to the patient, the last can respond "not applicable."

CONTACTS AND LOCATIONS:
Overall Officials: riccardo ruisi, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heyberger C, Auberger G, Babinet A, Anract P, Biau DJ. Patients with Revision Modern Megaprostheses of the Distal Femur Have Improved Disease-Specific and Health-Related Outcomes Compared to Those with Primary Replacements. J Knee Surg. 2018 Oct;31(9):822-826. doi: 10.1055/s-0037-1615298. Epub 2017 Dec 21. PMID 29270950
- [Background] Sadykova LR, Ntekim AI, Muyangwa-Semenova M, Rutland CS, Jeyapalan JN, Blatt N, Rizvanov AA. Epidemiology and Risk Factors of Osteosarcoma. Cancer Invest. 2020 May;38(5):259-269. doi: 10.1080/07357907.2020.1768401. Epub 2020 Jun 1. PMID 32400205
- [Background] Punzalan M, Hyden G. The role of physical therapy and occupational therapy in the rehabilitation of pediatric and adolescent patients with osteosarcoma. Cancer Treat Res. 2009;152:367-84. doi: 10.1007/978-1-4419-0284-9_20. PMID 20213402
- [Background] Kim TWB, Kumar RJ, Gilrain KL, Kubat E, Devlin C, Honeywell S, Amin SJ, Gutowski CJ. Team Approach: Rehabilitation Strategies for Patients After Osteosarcoma Reconstructive Surgery. JBJS Rev. 2020 Oct;8(10):e19.00225. doi: 10.2106/JBJS.RVW.19.00225. PMID 33044254
- [Background] Bekkering WP, Vliet Vlieland TP, Koopman HM, Schaap GR, Beishuizen A, Anninga JK, Wolterbeek R, Nelissen RG, Taminiau AH. A prospective study on quality of life and functional outcome in children and adolescents after malignant bone tumor surgery. Pediatr Blood Cancer. 2012 Jun;58(6):978-85. doi: 10.1002/pbc.23328. Epub 2011 Oct 11. PMID 21990185
- [Background] den Hollander D, Van der Graaf WTA, Fiore M, Kasper B, Singer S, Desar IME, Husson O. Unravelling the heterogeneity of soft tissue and bone sarcoma patients' health-related quality of life: a systematic literature review with focus on tumour location. ESMO Open. 2020 Oct;5(5):e000914. doi: 10.1136/esmoopen-2020-000914. PMID 33082266
- [Background] Ottaviani G, Robert RS, Huh WW, Jaffe N. Functional, psychosocial and professional outcomes in long-term survivors of lower-extremity osteosarcomas: amputation versus limb salvage. Cancer Treat Res. 2009;152:421-36. doi: 10.1007/978-1-4419-0284-9_23. PMID 20213405
- [Background] Robert RS, Ottaviani G, Huh WW, Palla S, Jaffe N. Psychosocial and functional outcomes in long-term survivors of osteosarcoma: a comparison of limb-salvage surgery and amputation. Pediatr Blood Cancer. 2010 Jul 1;54(7):990-9. doi: 10.1002/pbc.22419. PMID 20135700
- [Background] Bekkering WP, van Egmond-van Dam JC, Bramer JAM, Beishuizen A, Fiocco M, Dijkstra PDS. Quality of life after bone sarcoma surgery around the knee: A long-term follow-up study. Eur J Cancer Care (Engl). 2017 Jul;26(4). doi: 10.1111/ecc.12603. Epub 2016 Nov 7. PMID 28657211
- [Background] Eiser C. Assessment of health-related quality of life after bone cancer in young people: easier said than done. Eur J Cancer. 2009 Jul;45(10):1744-7. doi: 10.1016/j.ejca.2009.02.025. Epub 2009 Mar 25. PMID 19327986
- [Background] Bekkering WP, Vliet Vlieland TP, Koopman HM, Schaap GR, Schreuder HW, Beishuizen A, Tissing WJ, Hoogerbrugge PM, Anninga JK, Taminiau AH. Quality of life in young patients after bone tumor surgery around the knee joint and comparison with healthy controls. Pediatr Blood Cancer. 2010 May;54(5):738-45. doi: 10.1002/pbc.22439. PMID 20127850
- [Background] Taylor MF, Pooley JA. Sarcoma survivors' perspectives on their body image and functional quality of life post-resection/limb salvage surgery. Eur J Cancer Care (Engl). 2017 Nov;26(6). doi: 10.1111/ecc.12667. Epub 2017 Feb 21. PMID 28220660
- [Background] Bekkering WP, Billing L, Grimer RJ, Vlieland TP, Koopman HM, Nelissen RG, Taminiau AH. Translation and preliminary validation of the English version of the DUX questionnaire for lower extremity bone tumor patients (Bt-DUX): a disease-specific measure for quality of life. J Surg Oncol. 2013 Mar;107(4):353-9. doi: 10.1002/jso.23218. Epub 2012 Jul 17. PMID 22806913
- [Background] Barrera M, Teall T, Barr R, Silva M, Greenberg M. Health related quality of life in adolescent and young adult survivors of lower extremity bone tumors. Pediatr Blood Cancer. 2012 Feb;58(2):265-73. doi: 10.1002/pbc.23017. Epub 2011 Feb 11. PMID 21319288
- [Background] Liu Y, Hu A, Zhang M, Shi C, Zhang X, Zhang J. Correlation between functional status and quality of life after surgery in patients with primary malignant bone tumor of the lower extremities. Orthop Nurs. 2014 May-Jun;33(3):163-70. doi: 10.1097/NOR.0000000000000050. PMID 24845842
- [Background] Morri M, Bekkering PW, Cotti M, Meneghini M, Venturini E, Longhi A, Mariani E, Forni C. Cross-Cultural Validation of the Italian Version of the Bt-DUX: A Subjective Measure of Health-Related Quality of Life in Patients Who Underwent Surgery for Lower Extremity Malignant Bone Tumour. Cancers (Basel). 2020 Jul 23;12(8):2015. doi: 10.3390/cancers12082015. PMID 32717924
- [Background] Rossi L, Boffano M, Comandone A, Ferro A, Grignani G, Linari A, Pellegrino P, Piana R, Ratto N, Davis AM. Validation process of Toronto Exremity Salvage Score in Italian: A quality of life measure for patients with extremity bone and soft tissue tumors. J Surg Oncol. 2020 Mar;121(4):630-637. doi: 10.1002/jso.25849. Epub 2020 Jan 19. PMID 31957034
- [Background] Dong S, Sun K, Xie L, Xu J, Sun X, Ren T, Huang Y, Yang R, Tang X, Yang F, Gu J, Guo W. Quality of life and Q-TWiST were not adversely affected in Ewing sarcoma patients treated with combined anlotinib, irinotecan, and vincristine: (Peking University People's Hospital Ewing sarcoma trial-02, PKUPH-EWS-02). Medicine (Baltimore). 2021 Dec 23;100(51):e28078. doi: 10.1097/MD.0000000000028078. PMID 34941047
- [Background] Solooki S, Mostafavizadeh Ardestani SM, Mahdaviazad H, Kardeh B. Function and quality of life among primary osteosarcoma survivors in Iran: amputation versus limb salvage. Musculoskelet Surg. 2018 Aug;102(2):147-151. doi: 10.1007/s12306-017-0511-y. Epub 2017 Oct 13. PMID 29030830
- [Background] Bishop MW, Advani SM, Villarroel M, Billups CA, Navid F, Rivera C, Quintana JA, Gattuso JS, Hinds PS, Daw NC. Health-Related Quality of Life and Survival Outcomes of Pediatric Patients With Nonmetastatic Osteosarcoma Treated in Countries With Different Resources. J Glob Oncol. 2018 Sep;4:1-11. doi: 10.1200/JGO.2016.005967. Epub 2017 Mar 24. PMID 30241221
- [Background] Weschenfelder W, Gast-Froehlich S, Spiegel C, Vogt M, Hofmann GO. Factors influencing quality of life, function, reintegration and participation after musculoskeletal tumour operations. BMC Cancer. 2020 Apr 25;20(1):351. doi: 10.1186/s12885-020-06837-x. PMID 32334563